CLINICAL TRIAL: NCT00370071
Title: Open Label Study to Evaluate the Effect, Safety and Tolerability of 250µg (8 MIU) Interferon Beta 1b (Betaferon) Given Subcutaneously Every Other Day (for 24 Weeks) in Patients of Chinese Origin With Multiple Sclerosis
Brief Title: Open Label Study to Evaluate Effect, Safety and Tolerability of Betaferon Standard Dose of 250µg in Patients of Chinese Origin With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91386; MP-00102 (Other: Company internal); 308720 (Other: Company internal); 2014-004613-93 (EudraCT Number)
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon beta-1b (Betaseron, BAY86-5046) (Experimental): Interferon beta-1b 250 μg (8 MIU) subcutaneously (sc) every other day (e.o.d.)
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Interferon beta-1b 250 μg (8 MIU) subcutaneously (sc) every other day (e.o.d.)

SUMMARY:
The purpose of this study is to determine if the study drug is effective and safe in the treatment of Multiple Sclerosis (MS) in patients of Chinese origin.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany.

Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin
* diagnosis of Relapsing remitting multiple sclerosis or secondary progressive multiple sclerosis

Exclusion Criteria:

* Any disease other than Multiple Sclerosis (MS) that could better explain the patients signs and symptoms
* HIV (human immunodeficiency virus) infections
* Hepatitis A
* Syphilis
* immunodeficiency
* rheumatic disease or Sjogren syndrome
* heart disease
* severe depression
* pregnancy or lactation
* conditions interfering with Magnetic Resonance Imaging (MRI)
* Gadolinium DTPA (Gadovist, contrast agent) allergy
* allergy against human proteins, paracetamol, acetaminophen and ibuprofen intolerance
* participation in other trial

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- China (2):
  - Beijing
  - Shanghai

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in China between 08 November 2006 (first subject first visit) and 26 September 2008 (last subject last visit).
Pre-assignment Details: After a 3-month pre-treatment period with no MS-specific treatment, 39 subjects entered the 6-month treatment period. Of the 84 subjects screened, 40 subjects did not meet the inclusion/exclusion criteria, 3 subjects withdrew their consent, and 2 subjects died during pre-treatment.
Period: Overall Study
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Started | 39
Completed | 37
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Interferon Beta-1b (Betaseron, BAY86-5046): Interferon beta-1b 250 micrograms (8 MIU [million international units]) subcutaneously every other day.
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Full Range); unit: years] | 31.6 [17 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 13
Gadolinium enhancing lesions (T1) at screening [Number; unit: participants]
  no lesions | 5
  1-3 lesions | 23
  >= 4 lesions | 11
Type of Multiple Sclerosis [Number; unit: participants]
  Relapsing-remitting (RR) | 36
  Secondary progressive (SP) | 3
Expanded disability status scale at screening (EDSS) [Mean (Full Range); unit: Points on a scale] — The EDSS is a scale based on the standardized neurological examination which comprised of optic, brain stem/cranial nerves, pyramidal, cerebellar, sensory, vegetative, and cerebral functions, as well as walking ability. The EDSS scores range from 0.0 (normal) to 10.0 (dead). A score of 2 to 3 indicates minimal to moderate disability.
  Points on a scale | 2.26 [0 to 5.0]
New Gd-enhancing lesions during 3-month pre-treatment [Mean (Standard Deviation); unit: lesions] | 2.6 (4.1)
New or enlarging T2 lesions during 3-month pre-treatment [Mean (Standard Deviation); unit: lesions] | 2.2 (3.2)
Newly active lesions during 3-month pre-treatment [Mean (Standard Deviation); unit: lesions] | 4.8 (7.1)
Previous Multiple Sclerosis relapses [Mean (Standard Deviation); unit: relapses] | 2.8 (1.7)
T2 lesions at screening [Mean (Standard Deviation); unit: lesions] | 45.1 (32.9)
Time since onset of Multiple Sclerosis [Mean (Standard Deviation); unit: years] | 3.5 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Number of Newly Active Lesions in Magnetic Resonance Imaging (MRI) Per Three Months During the 6-month Treatment Period and the Number of Newly Active Lesions During 3-month Pre-treatment
Description: The primary efficacy variable was calculated by subtracting the number of newly active lesions during the 3-month pre-treatment period from the cumulative number of newly active lesions during the 6-month treatment period divided by 2 (number of newly active lesions per three months, new lesion frequency per 3 months)
Time Frame: after 6 months of treatment as compared to 3-month pre-treatment
Population: The primary analysis set included all MRS (MRI set) patients who had at least one dose of study drug and at least one evaluable post-baseline MRI scan. The primary endpoint data was missing for one patient.
Measure: Median (Full Range); unit: lesions
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 38
lesions | -1.5 [-35 to 6.5]
Statistical Analysis 1: Comparison: Interferon Beta-1b (Betaseron, BAY86-5046); In this single arm study, the number of newly active lesions per 3 months during treatment was compared to the number of newly active lesions during 3-month pre-treatment (Alternative hypothesis: Number of lesions is reduced during treatment with Interferon beta-1b). The sample size was calculated for the use of the one-sided Wilcoxon-Signed-Rank test at level 2.5% (Power of 90% - anticipating P(X<Y)=0.15 and allowing for 25% exclusion from Per Protocol Set); Test type: Superiority or Other; p < 0.0001, Wilcoxon-Signed-Rank test — one-sided p-value (one-sided test level 2.5%)

2. Secondary Outcome: Difference Between the Number of New Gadolinium (Gd)-Enhancing Lesions Per 3 Months During the 6-month Treatment Period and the Number of New Gd-enhancing Lesions During 3-month Pre-treatment
Description: This secondary endpoint (component of the primary endpoint) was calculated by subtracting the number of new Gd-enhancing lesions during the 3-month pre-treatment period from the cumulative number of new Gd-enhancing lesions during the 6-month treatment period divided by 2 (number of new Gd-enhancing lesions per three months)
Time Frame: after 6 months of treatment as compared to 3-month pre-treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: lesions
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 38
lesions | -0.5 [-22 to 1.5]
Statistical Analysis 1: Comparison: Interferon Beta-1b (Betaseron, BAY86-5046); Test type: Superiority or Other; p < 0.0001, Wilcoxon-Signed-Rank test — one-sided p-value (one-sided test level 2.5%)

3. Secondary Outcome: Difference Between the Number of New or Enlarging T2 Lesions Per 3 Months During the 6-month Treatment Period and the Number of New or Enlarging T2 Lesions During 3-month Pre-treatment
Description: This secondary endpoint (component of the primary endpoint) was calculated by subtracting the number of new or enlarging T2 lesions during the 3-month pre-treatment period from the cumulative number of new or enlarging T2 lesions during the 6-month treatment period divided by 2 (number of new T2 lesions per three months) based on non-enhancing lesions on T1 weighted scans
Time Frame: after 6 months of treatment as compared to the 3-month pre-treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: lesions
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 38
lesions | 0 [-13 to 6.5]
Statistical Analysis 1: Comparison: Interferon Beta-1b (Betaseron, BAY86-5046); Test type: Superiority or Other; p = 0.0017, Wilcoxon-Signed-Rank test — one-sided p-value (one-sided test level 2.5%)

4. Secondary Outcome: Volume of Gadolinium-enhancing Lesions at Baseline, Weeks 12 and 24
Description: In the categories listed below, "N" signifies the number of subjects evaluable for the timepoints.
Time Frame: Baseline, Weeks 12 and 24
Population: MRS
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
cubic millimeter (mm^3)
  Baseline (N=39) | 585 (869)
  Week 12 (N=38) | 93 (184)
  Week 24 (N=37) | 648 (2788)
Statistical Analysis 1: Comparison: Interferon Beta-1b (Betaseron, BAY86-5046); Lesion volume at Week 12. 38 subjects were evaluated; Test type: Superiority or Other; p < 0.0001, Wilcoxon-Signed-Rank test; One-sided p-value from Wilcoxon-Signed-Rank-Test for comparing the baseline visit to treatment visits
Statistical Analysis 2: Comparison: Interferon Beta-1b (Betaseron, BAY86-5046); Lesion volume at Week 24. 37 subjects were evaluated; Test type: Superiority or Other; p = 0.0019, Wilcoxon-Signed-Rank test

5. Secondary Outcome: Number of New Gadolinium (T1)-Enhancing Lesions at Baseline, Weeks 12 and 24
Description: In the categories listed below, "N" signifies the number of subjects evaluable for the timepoints.
Time Frame: Baseline, Weeks 12 and 24
Population: MRS
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
Lesions
  Baseline (N=39) | 2.8 (4.15)
  Week 12 (N=38) | 0.5 (1.01)
  Week 24 (N=37) | 0.8 (1.83)

6. Secondary Outcome: Number of T2 Lesions at Baseline, Weeks 12 and 24
Description: In the categories listed below, "N" signifies the number of subjects evaluable for the timepoints.
Time Frame: Baseline, Weeks 12 and 24
Population: MRS
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
Lesions
  Baseline (N=39) | 48.7 (35.77)
  Week 12 (N=38) | 48.8 (35.21)
  Week 24 (N=37) | 44.6 (31.54)

7. Secondary Outcome: Assessment of Relapses: Relapse Rate
Description: A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical event. The abnormality must be present for at least 24 hours and occur in the absence of fever (axillary temperature more than (>) 37.5 degree celsius / 99.5 degree fahrenheit) or known infection. A relapse must be confirmed by a documented report from a physician or by objective assessment. The relapse rate was calculated on an annualized basis. Annualized relapse rate is the average number of relapses in a year calculated by negative binomial regression as the sum of confirmed relapses of all subjects in the group divided by the sum of the number of days on study of all subjects in the group and multiplied by 365.25.
Time Frame: Baseline up to Week 24
Population: Full analysis set (FAS)
Measure: Number; unit: relapses per year
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
relapses per year | 0.38

8. Secondary Outcome: Assessment of Relapses: Number of Relapses
Description: A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical event. The abnormality must be present for at least 24 hours and occur in the absence of fever (axillary temperature >37.5 degree celsius / 99.5 degree fahrenheit) or known infection. A relapse must be confirmed by a documented report from a physician or by objective assessment. In the categories listed below, "N" signifies the number of subjects evaluable for the timepoints, and same subjects were counted more than once under each category.
Time Frame: 3 and 6 months
Population: FAS with all subjects who had reported relapses
Measure: Number; unit: relapses
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 10
relapses
  3 months (N=6) | 6
  6 months (N=6) | 7

9. Secondary Outcome: Assessment of Relapses: Percentage of Relapse-free Subjects After 24 Weeks
Description: A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical event. The abnormality must be present for at least 24 hours and occur in the absence of fever (axillary temperature >37.5 degree celsius / 99.5 degree fahrenheit) or known infection. A relapse must be confirmed by a documented report from a physician or by objective assessment.
Time Frame: After 24 weeks
Population: FAS
Measure: Number; unit: percentage of subjects
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
percentage of subjects | 84.6

10. Secondary Outcome: Assessment of Relapses: Relapse Severity
Description: A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical event. The abnormality must be present for at least 24 hours and occur in the absence of fever (axillary temperature >37.5 degree celsius / 99.5 degree fahrenheit) or known infection. A relapse must be confirmed by a documented report from a physician or by objective assessment. A major relapse was defined based on changes on EDSS with the following additional criteria to be met: objective neurological impairment, correlating with the subject's reported symptoms, defined as either increase in at least one of the functional systems of the EDSS score or increase of the total EDSS score. Relapses which did not meet the criteria of major relapses were considered as non-major.
Time Frame: Baseline up to Week 24
Population: FAS with all subjects who had reported relapses
Measure: Number; unit: relapses
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 10
relapses
  Major | 1
  Non-major | 12

11. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: The EDSS is a scale based on the standardized neurological examination which comprised of optic, brain stem/cranial nerves, pyramidal, cerebellar, sensory, vegetative, and cerebral functions, as well as walking ability. The EDSS scores range from 0.0 (normal) to 10.0 (dead). A score of 2 to 3 indicates minimal to moderate disability.
Time Frame: Pre-treatment on Day 1, Week 24
Population: FAS subjects with EDSS assessments at the end of the study (Week 24)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 37
Scores on a scale
  Pre-treatment | 2.06 (1.6)
  Week 24 | 1.81 (1.72)

12. Secondary Outcome: Percentage of Subjects Without EDSS Progression
Description: The EDSS is a scale based on the standardized neurological examination which comprised of optic, brain stem/cranial nerves, pyramidal, cerebellar, sensory, vegetative, and cerebral functions, as well as walking ability.The EDSS scores range from 0.0 (normal) to 10.0 (dead). A score of 2 to 3 indicates minimal to moderate disability. An EDSS progression was defined as increase in EDSS greater than or equal to (>=) 1.0 points (in the treatment period as compared to baseline).
Time Frame: Baseline up to Week 24
Population: FAS
Measure: Number; unit: percentage of subjects
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Number analyzed (Participants) | 39
percentage of subjects | 87.2

ADVERSE EVENTS:
Time Frame: Baseline up to the end of the study (Week 24)
Description: Treatment-emergent adverse events were defined as adverse events which were not recorded before the start of study treatment or, if pre-existent, had increased in intensity after the start of study treatment.
Arm/Group | Interferon Beta-1b (Betaseron, BAY86-5046)
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 34/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1b (Betaseron, BAY86-5046) (N=39)
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye movement disorder (Eye disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatique (General disorders) | 3
Influenza like illness (General disorders) | 16
Injection site erythema (General disorders) | 3
Injection site pain (General disorders) | 4
Injection site reaction (General disorders) | 3
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Hepathic function abnormal (Hepatobiliary disorders) | 7
Nasopharyngitis (Infections and infestations) | 3
Fibula fracture (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2
white blood cell count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Facial palsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Menstruation delayed (Reproductive system and breast disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less